CLINICAL TRIAL: NCT03705884
Title: Molecular Imaging in Cardiovascular Disease Using Hybrid Positron Emission Tomography/Magnetic Resonance Imaging (PET/MR): Cardiac Sarcoidosis
Brief Title: PET/MR Imaging In Patients With Cardiac Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AC17010
Record Dates: First submitted 2018-08-08; First posted 2018-10-15 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Sarcoidosis
MeSH Terms: interventions — Fluorodeoxyglucose F18; Prednisolone

STUDY DESIGN:
Intervention Model Description: Patients and healthy subjects will be allocated in a non-randomised fashion to either corticosteroid or control arms, for parallel comparison within the two groups. The corticosteroid is recognised treatment for the condition and is being used to observe the impact on diagnostic imaging; no treatment effects are being studied or are endpoints of the study (i.e. the study is not a clinical trial of treatment in cardiac sarcoidosis with corticosteroid).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Sarcoidosis (Other): Patients with an established diagnosis of cardiac sarcoidosis.
  Interventions: Other: 18F-FDG; Drug: Prednisolone
- Healthy volunteers (Other): Healthy volunteer subjects of similar age and gender to patient cohort.
  Interventions: Other: 18F-FDG; Drug: Prednisolone

INTERVENTIONS:
Other: 18F-FDG — Hybrid 18F-FDG PET/MR imaging for observational diagnostic purposes.
Drug: Prednisolone — Oral course of Prednisolone for treatment of sarcoidosis (patient cohort) or as control (healthy volunteer cohort)

SUMMARY:
PET scanning (positron emission tomography) is a well-established technique used to identify areas of interest within the body. It involves injecting a radioactive tracer which highlights abnormal areas. It has recently been combined with CT (computed tomography) and MRI (magnetic resonance imaging) scanning to more accurately identify abnormalities within the heart. Cardiac sarcoidosis, a condition which causes scarring and inflammation within the heart muscle, is of particular interest.

The study makes use of hybrid PET/MR scanning using a designated scanner which enables PET scanning combined with MRI scanning. This will allow imaging of abnormal areas within the heart in this condition alongside treatment regimens in a way which hasn't been done before. If successful, this imaging method will play a key role in diagnosing, quantifying and monitoring these conditions.

All participants will undergo PET scanning, where a radioactive tracer is injected into a vein before the scan. The radioactive substance only lasts for a short time and is safe, passed out of the body in urine. The scan will be performed twice; once before treatment and once after treatment has been established. A cohort of healthy volunteers will undergo scanning in exactly the same way to enable us to compare the results with hearts of people who don't have cardiac sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

Cardiac Sarcoidosis Patients:

* Aged over 40 years
* Completion of informed consent
* Established diagnosis of cardiac sarcoidosis
* Established diagnosis as per HRS recommended diagnostic criteria

Healthy Volunteers:

* Aged over 40
* Completion of informed consent

Exclusion Criteria:

* All participants:
* Inability or unwilling to give informed consent
* Women who are pregnant, breastfeeding or of child-bearing potential (women who have experienced menarche, are pre-menopausal and have not been sterilised) will not be enrolled into the trial.
* Major intercurrent illness with life-expectancy <2 years.
* Renal dysfunction (eGFR less than or equal to 30ml/min/1.73m2)
* Adverse reaction or hypersensitivity to 18F-FDG PET tracer
* NYHA Class IV heart failure
* Patients with atrial fibrillation and poor rate control
* Contraindications to MRI scanning
* Previous history of contrast allergy of adverse reactions (Gadolinium-containing agents)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Myocardial 18F-FDG uptake | Within 1 year
  Quantification of myocardial PET tracer uptake before steroid therapy
Myocardial 18F-FDG uptake | Within 1 year
  Quantification of myocardial PET tracer uptake after steroid therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marc R Dweck, MD PhD, Study Director — University of Edinburgh
Locations (1):
- Queen's Medical Research Institute, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No